CLINICAL TRIAL: NCT04828369
Title: Efficacy and Safety of EUS-Guided Coil Embolization Combined With Endoscopic Cyanoacrylate Injection Versus Balloon-Occluded Retrograde Transvenous Obliteration for Gastric Varices With High-risk Ectopic Embolism
Brief Title: Efficacy and Safety of EUS-Guided Therapy Versus BRTO for Gastric Varices With Shunt
Status: Completed | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, ChenMingkai, Professor, Renmin Hospital of Wuhan University
Other Study IDs: 2021F024
Record Dates: First submitted 2021-03-25; First posted 2021-04-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Portal Hypertension; Liver Cirrhosis; Gastric Varix; Portosystemic Shunt
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis; Esophageal and Gastric Varices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EUS group: Patients who received EUS-guided coil embolization combined with endoscopic cyanoacrylate injection
  Interventions: Procedure: EUS-guided coil embolization combined with endoscopic cyanoacrylate injection
- BRTO group: Patients who received balloon-occluded retrograde transvenous obliteration (BRTO)
  Interventions: Procedure: balloon-occluded retrograde transvenous obliteration

INTERVENTIONS:
Procedure: EUS-guided coil embolization combined with endoscopic cyanoacrylate injection — (1) Standard diagnostic endoscopy was first performed. Fundal varices were assessed using the classification of Sarin's. (2) intraluminal water filling of the gastric fundus to use EUS to assess the anatomy of gastric varices, observe the blood flow, scan the portal venous system, left renal vein, confirm the location of the shunt, and measure the diameter of the shunt. (3) Punctured the gastric fundal variceal vein at the lower esophagus near the cardia and placed the coil into the shunt and immediately injected with sclerosant and cyanoacrylate under the guidance of EUS. (4) Sclerosant and cyanoacrylate were injected into the gastric fundal varices by a sandwich method (cyanoacrylate, sclerosant and cyanoacrylate) via endoscope. (5) After the injection, use color Doppler ultrasound to observe the blood flow in the variceal veins to evaluate the embolization effect.
  Groups: EUS group
Procedure: balloon-occluded retrograde transvenous obliteration — (1)A balloon occlusive catheter was inserted into the shunt via the right femoral vein. (2)Investigators performed angiography to evaluate the size and location of GV and the shunt during balloon occlusion. Shunt was occluded by Fogarty balloon. The diameter of the balloon was chosen according to the diameter of shunt. (3)Then investigators injected sclerosant into the portosystemic shunt. (4)Finally, the balloon left in place for 24 hours was gradually deflated when complete occlusion of blood flow of the target shunt was achieved.
  Groups: BRTO group

SUMMARY:
This study is a retrospective, multi-center and observational clinical study. Renmin Hospital of Wuhan University, Beijing Friendship Hospital, Capital Medical University, The fifth medical center of PLA General Hospital, Zhongshan Hospital, Fudan University, Shanghai, Nanjing Drum Tower Hospital affiliated Nanjing University Medical School and Xiangyang Central Hospital will participate in the study. Investigators would like to provide evidence-based medical evidence by evaluating and comparing the efficacy and safety of endoscopic ultrasound (EUS)-guided coil embolization combined with endoscopic cyanoacrylate injection and balloon-occluded retrograde transvenous obliteration (BRTO) in the treatment of gastric varices (GV) with spontaneous portosystemic shunt (SPSS).

Between January 2014 and December 2020, patients with GV secondary to portal hypertension admitted to a tertiary medical center, are enrolled consecutively according to the following criteria: (1) age≥18 years; (2)endoscopic examination confirms the presence of GV; (3) CTA of the portal system and EUS revealed the presence of SPSS, the diameter was between 5 mm to 15 mm; (4) treatment with EUS-guided coil combined with endoscopic cyanoacrylate injection or BRTO. Exclusion criteria are as follows: (1)malignant tumors; (2) hepatic encephalopathy, hepatorenal syndrome or multiple organ failure; (3) previously received esophagus or stomach surgery; (4) pregnant.

Investigators will collect patients' data of baseline character, treatment, postoperative and follow-up. All patients will be followed up until the progress of the disease or the end of the study. And rebleeding, ectopic embolism, survival, and sequential treatment will be recorded during the follow-up period.

The primary endpoint are five-day rebleeding rate and six-week mortality rate. The secondary endpoint are: technical success rate, incidence of ectopic embolism, eradication of GV, one-year rebleeding rate, one-year mortality rate, and cost-effectiveness ratio. All data and information use SPSS statistical software to complete all statistical analysis.

DETAILED DESCRIPTION:
Because the efficacy and safety of EUS-guided coil embolization combined with endoscopic cyanoacrylate injection and BRTO in the treatment of GV with SPSS have different conclusions in different studies. Investigators based on that the five-day rebleeding rate of EUS-guided coil embolization combined with endoscopic cyanoacrylate injection is 7%, BRTO is 10%. The number of people in the two groups are equal, significant level (α) is 0.05, and the test power is 0.8. Each group requires 35 patients. Because of the 10% loss to follow-up, the sample capacity is 39.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years
* endoscopic examination confirmed the presence of gastric varices
* CTA of the portal system and EUS revealed the presence of spontaneous portosystemic shunt (SPSS) that the diameter was between 5 mm to 15 mm
* treatment with EUS-guided coil combined with endoscopic cyanoacrylate injection or BRTO

Exclusion Criteria:

* malignant tumors
* hepatic encephalopathy, hepatorenal syndrome or multiple organ failure
* previously received esophagus or stomach surgery
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects in this study are patients with gastric varices resulted from portal hypertension. And the presence of spontaneous portosystemic shunt has been confirmed by CTA or EUS.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
five-day rebleeding rate | 5 days after treatment
  Rebleeding is defined as recurrent melena or hematemesis and is evaluated via endoscopy when possible.
six-week mortality rate | 6 weeks after treatment
  Patients died in six weeks after treatment due to all causes.

SECONDARY OUTCOMES:
technical success rate | in the procedure of treatment
  The coil or balloon was successfully employed and occluded the shunt
incidence of ectopic embolism | up to 3 years after treatment
  Patients occurred ectopic embolism after treatment confirmed by CTA, ultrasound, etc, with or without clinical manifestation
eradication of gastric varices | 1 year after treatment
  Eradication of the gastric varices is defined as absence of gastric varices on endoscopy or absence of blood flow of gastric varices on endoscopic ultrasound
one-year rebleeding rate | 1 year after treatment
  Rebleeding is defined as recurrent melena or hematemesis and is evaluated via endoscopy when possible
one-year mortality rate | 1 year after treatment
  Patients died in one year after treatment due to all causes.

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Chen, PHD, Study Director — Renmin Hospital of Wuhan University
Locations (1):
- Mingkai Chen, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Boregowda U, Umapathy C, Halim N, Desai M, Nanjappa A, Arekapudi S, Theethira T, Wong H, Roytman M, Saligram S. Update on the management of gastrointestinal varices. World J Gastrointest Pharmacol Ther. 2019 Jan 21;10(1):1-21. doi: 10.4292/wjgpt.v10.i1.1. PMID 30697445
- [Result] Wu Q, Shen L, Chu J, Ma X, Jin B, Meng F, Chen J, Wang Y, Wu L, Han J, Zhang W, Ma W, Wang H, Li H. Characterization of uncommon portosystemic collateral circulations in patients with hepatic cirrhosis. Oncol Lett. 2015 Jan;9(1):347-350. doi: 10.3892/ol.2014.2626. Epub 2014 Oct 22. PMID 25435990
- [Result] Qi X, Qi X, Zhang Y, Shao X, Wu C, Wang Y, Wang R, Zhang X, Deng H, Hou F, Li J, Guo X. Prevalence and Clinical Characteristics of Spontaneous Splenorenal Shunt in Liver Cirrhosis: A Retrospective Observational Study Based on Contrast-Enhanced Computed Tomography (CT) and Magnetic Resonance Imaging (MRI) Scans. Med Sci Monit. 2017 May 25;23:2527-2534. doi: 10.12659/msm.901656. PMID 28542116
- [Result] Zardi EM, Uwechie V, Caccavo D, Pellegrino NM, Cacciapaglia F, Di Matteo F, Dobrina A, Laghi V, Afeltra A. Portosystemic shunts in a large cohort of patients with liver cirrhosis: detection rate and clinical relevance. J Gastroenterol. 2009;44(1):76-83. doi: 10.1007/s00535-008-2279-1. Epub 2009 Jan 22. PMID 19159076
- [Result] von Herbay A, Frieling T, Haussinger D. Color Doppler sonographic evaluation of spontaneous portosystemic shunts and inversion of portal venous flow in patients with cirrhosis. J Clin Ultrasound. 2000 Sep;28(7):332-9. doi: 10.1002/1097-0096(200009)28:73.0.co;2-9. PMID 10934332
- [Result] Park JK, Saab S, Kee ST, Busuttil RW, Kim HJ, Durazo F, Cho SK, Lee EW. Balloon-Occluded Retrograde Transvenous Obliteration (BRTO) for Treatment of Gastric Varices: Review and Meta-Analysis. Dig Dis Sci. 2015 Jun;60(6):1543-53. doi: 10.1007/s10620-014-3485-8. Epub 2014 Dec 18. PMID 25519690
- [Result] Garcia-Tsao G, Abraldes JG, Berzigotti A, Bosch J. Portal hypertensive bleeding in cirrhosis: Risk stratification, diagnosis, and management: 2016 practice guidance by the American Association for the study of liver diseases. Hepatology. 2017 Jan;65(1):310-335. doi: 10.1002/hep.28906. Epub 2016 Dec 1. No abstract available. PMID 27786365
- [Result] Mohan BP, Chandan S, Khan SR, Kassab LL, Trakroo S, Ponnada S, Asokkumar R, Adler DG. Efficacy and safety of endoscopic ultrasound-guided therapy versus direct endoscopic glue injection therapy for gastric varices: systematic review and meta-analysis. Endoscopy. 2020 Apr;52(4):259-267. doi: 10.1055/a-1098-1817. Epub 2020 Feb 6. PMID 32028533